CLINICAL TRIAL: NCT02327455
Title: Integrated RF and B-mode Deformation Analysis for 4D Stress Echocardiography
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was never started.
Sponsor: Yale University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1406014091; R01HL0121226 (Other Grant/Funding Number: NHLBI); 2R01HL121226-05A1 (NIH)
Record Dates: First submitted 2014-11-25; First posted 2014-12-30 (Estimated); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stress Dobutamine Echocardiographic 4DE Image System (Experimental): Subjects will undergo their clinically indicated stress dobutamine echocardiographic studies using our standard clinical graded dobutamine stress imaging protcol, employing the iE33 4DE system.
  Interventions: Procedure: Stress Dobutamine Echocardiographic using 4DE System

INTERVENTIONS:
Procedure: Stress Dobutamine Echocardiographic using 4DE System — Subjects will undergo their clinically indicated stress dobutamine echocardiographic studies using our standard clinical graded dobutamine stress imaging protcol, employing the iE33 4DE system.

SUMMARY:
The specific aim of this clinical trial is to translate the investigators new 4DE (three sptial dimensions pluse time) stress echocardiographic method to patients with coronary artery disease referred for clinically indicated dobutamine stress/rest echo to evaluate the reproducibility of the technique in this clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age, referred for clinically indicated dobutamine rest/stress TTE
* Provide written informed consent to participate in the study
* Availability for repease rest/stress TTE within on eweek of clinically indicated study

Exclusion Criteria:

* Unable to give informed consent
* Unstable hemodynamics that would not allow for repease rest/stress dobutamine transthoracic imaging
* Recurrent life threatening arrhythmias
* Heart rate >110 BPM
* Inadequate windows for transthoracic imagine
* Patients that have a narrow-angle glaucoma (contraindication for atropine)
* Change in cardiac medications or management including, coronary revascularization beween intial and repeat TTE study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-07 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Number of Subjects With an Interpretable 4DE Image | After Stress Echocardiography (Approximately 2 hours)
  This outcome will measure feasibility. Data from images will be analyzed with the integrated speckle/shape tracking approach (the method uses boundary detection/shape tracking to quantify left ventricular myocardial deformation)

CONTACTS AND LOCATIONS:
Overall Officials: Albert Sinusas, MD, Principal Investigator — Yale University